CLINICAL TRIAL: NCT04916444
Title: Dystonia Treatment With Injections Supplemented By Transcranial Magnetic Stimulation
Acronym: D-TWIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Dystonia Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202101156; OCR40846 (Other: UF OnCore)
Record Dates: First submitted 2021-05-20; First posted 2021-06-07 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Cervical Dystonia
Keywords: rTMS; cervical dystonia; botulinum toxin
MeSH Terms: conditions — Torticollis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients were randomized to one of two conditions during session 1: active or sham rTMS. During session 2, patients underwent whichever condition they did not undergo in session 1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A sham coil was used for sham rTMS. Both conditions underwent the exact same study procedures except the sham coil did not deliver pulses; it did still deliver a sound and tapping sensation meant to mimic the real rTMS coil, but no real stimulation was provided in this condition. Patients and outcomes assessors were not made aware of the condition that the participant was partaking in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active rTMS (Active Comparator): Active rTMS will use a figure of eight TMS coil that will deliver real neurostimulation pulses to the patients.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham rTMS will use a sham figure of eight TMS coil that sounds and looks like a real rTMS coil, except no neurostimulation is being delivered to the patient.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — repetitive transcranial magnetic stimulation is a painless, noninvasive form of neurostimulation. This study uses an accelerated protocol in which the neurostimulation pulses are delivered in 4 sessions per day over 4 consecutive days (16 total sessions). Active or sham rTMS will be provided at 9 weeks following botox injections.
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
We applied 16 sessions of rTMS over 4 consecutive days for adult patients suffering from cervical dystonia who received botulinum toxin (BoNT) injections on a regular basis. The TMS protocol took place 9 weeks following their last BoNT injection. The primary outcome measure was improvement in cervical dystonia as measured by the TWSTRS scale. The secondary outcome measures included mood, cognition, and gait measures.

DETAILED DESCRIPTION:
This was a crossover study design in which patients were randomized to active or sham stimulation during session 1 (S1) and then crossed over to the condition they were not randomized to at first during session 2 (S1). Patients who were receiving BoNT injections for cervical dystonia on a regular basis but only noted benefit from BoNT for 9 weeks or less were eligible to participate. The total study protocol took place over 24 weeks. During week 1, patients had their regularly scheduled botox injections. During week 9, patients underwent either active or sham rTMS, as detailed below. They had outcome measures obtained at week 9 (S1:T0; baseline/pre-TMS), week 10 (S1:T1; post-TMS), and week 12 (S1:T2; 2 weeks post-TMS). At week 12, they underwent their regularly scheduled BoNT injections. During week 21, patients underwent either active or sham rTMS, whichever condition they were not randomized into during the first session. They then had outcome measures obtained at week 21 (S2:T0; baseline/pre-TMS), week 22 (S2:T1; post-TMS), and week 24 (S2:T2; 2 weeks post-TMS).

The neurostimulation protocol was as follows: The dPMC target was defined as 1 cm medial and 2 cm anterior to the site of RMT acquisition. The rTMS protocol was as follows: each session consisted of 1-Hz rTMS over the dPMC for 30 minutes (1800 pulses) at 90% of the RMT. Patients received 4 sessions per day for 4 consecutive days with a 10-minute break between each session. The daily duration of the rTMS protocol, including breaks, lasted approximately 160 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-85 years of age who receive regular botulinum toxin (BoNT) scheduled every 12 weeks, on stable optimized doses but with reported benefits lasting ≤ 9 weeks for 2 consecutive cycles. Patents followed at our center routinely fill out a self-reported form to document the duration of benefits perceived with BoNT therapy. Participants will be allowed to continue oral medications that they are taking for dystonia concurrently but will not be allowed to change their concurrent medication regimen throughout the duration of the study.

Exclusion Criteria:

* Presence of metallic objects or neurostimulators in the brain
* Pregnancy
* History of active seizures or epilepsy
* Patients with severe scoliosis or other gait impairment that will preclude them from participating in gait evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yu, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, randomized, double-blind, crossover study. Five participants were recruited at the University of Florida Norman Fixel Institute for Neurological Diseases. Recruitment occurred between January and February 2022.
Pre-assignment Details: At 9 weeks after their regularly scheduled botulinum toxin injection visits, the participants were randomly assigned to receive either active rTMS first or sham first.
Groups:
- Active rTMS First: The active repetitive transcranial magnetic stimulation (rTMS) was provided at 9 weeks following the botulinum toxin injection.
  First, a clinical therapeutic NeuroStar TMS coil (Neuronetics, Malvern, PA) was used to determine the resting motor threshold (RMT), defined as the lowest stimulation intensity required to evoke a muscle twitch in a target muscle (first dorsal interosseus) for 5/10 pulses. The dPMC target was defined as 1 cm medial and 2 cm anterior to the site of RMT acquisition, consistent with how this target has been defined in the literature previously.
  Then, the clinical therapeutic TMS coil was switched to the active NeuroStar TMS coil. The rTMS protocol was as follows: each session consisted of 1-Hz rTMS over the dPMC for 30 minutes (1800 pulses) at 90% of the RMT. This study used an accelerated protocol: patients received 4 sessions per day for 4 consecutive days with a 10-minute break between each session. The daily duration of the rTMS protocol, including breaks, lasted approximately 160 minutes.
- Sham rTMS First: The sham rTMS was provided at 9 weeks following the botulinum toxin injection.
  First, the participants underwent the same procedure for identifying the target location and RMT as was used in patients receiving active rTMS.
  Then, the simulated rTMS was administered using a NeuroStar sham coil, which looked the same as the active stimulation coil and produced discharge noise and vibration without stimulating the cerebral cortex. This technique has been suggested to provide the most effective blinding compared to other methods used in randomized, controlled rTMS studies. The physician who set up the active and sham coils played no role in outcome measure assessments in order to maintain blinding.
Period: First Intervention (4 Days)
Arm/Group | Active rTMS First | Sham rTMS First
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Washout (12 Weeks)
Arm/Group | Active rTMS First | Sham rTMS First
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Second Intervention (4 Days)
Arm/Group | Active rTMS First | Sham rTMS First
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS First | Sham rTMS First | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 63.3 [52 to 71] | 76 [73 to 79] | 68.4 [52 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5
Duration since dystonia onset [Mean (Full Range); unit: years] | 11 [6 to 20] | 6.5 [5 to 8] | 9.2 [5 to 20]
Sensory trick [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2
  No | 1 | 2 | 3
Other dystonic features [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 2 | 2 | 4
Family history [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 3 | 2 | 5
Neurotoxin [Count of Participants; unit: Participants]
  OnabotulinumtoxinA | 3 | 0 | 3
  IncobotulinumtoxinA | 0 | 1 | 1
  RimabotulinumtoxinB | 0 | 1 | 1
Dosage [Mean (Full Range); unit: units] — Population: Out of the 5 participants, 3 were receiving onabotulinumtoxinA injection, 1 incobotulinumtoxinA injection, and 1 rimabotulinumtoxinB injection.
  units
    OnabotulinumtoxinA: number analyzed (Participants) | 3 | 0 | 3
    OnabotulinumtoxinA | 323.3 [220 to 400] |  | 323.3 [220 to 400]
    IncobotulinumtoxinA: number analyzed (Participants) | 0 | 1 | 1
    IncobotulinumtoxinA |  | 370 [370 to 370] | 370 [370 to 370]
    RimabotulinumtoxinB: number analyzed (Participants) | 0 | 1 | 1
    RimabotulinumtoxinB |  | 10000 [10000 to 10000] | 10000 [10000 to 10000]

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: This is an objective scale evaluating patients on a variety of features including maximal excursion, duration, effects of sensory trick, shoulder elevation, range of motion, and time. Scores range from 0 to 85 where a higher score indicates more severity.
Time Frame: Before rTMS (Session 1: Week 9, Session 2: Week 21), Immediately after rTMS (Session 1: Week 10, Session 2: Week 22), 2 weeks after rTMS (Session 1: Week 12, Session 2: Week 24)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active rTMS: Participants who received active repetitive transcranial magnetic stimulation (rTMS) during either the first intervention or the second intervention period.
  First, a clinical therapeutic NeuroStar TMS coil (Neuronetics, Malvern, PA) was used to determine the resting motor threshold (RMT), defined as the lowest stimulation intensity required to evoke a muscle twitch in a target muscle (first dorsal interosseus) for 5/10 pulses. The dPMC target was defined as 1 cm medial and 2 cm anterior to the site of RMT acquisition, consistent with how this target has been defined in the literature previously.
  Then, the clinical therapeutic TMS coil was switched to the active NeuroStar TMS coil. The rTMS protocol was as follows: each session consisted of 1-Hz rTMS over the dPMC for 30 minutes (1800 pulses) at 90% of the RMT. This study used an accelerated protocol: patients received 4 sessions per day for 4 consecutive days with a 10-minute break between each session. The daily duration of the rTMS protocol, including breaks, lasted approximately 160 minutes.
- Sham rTMS: Participants who received sham repetitive transcranial magnetic stimulation (rTMS) during either the first intervention or the second intervention period.
  First, the participants underwent the same procedure for identifying the target location and RMT as was used in patients receiving active rTMS.
  Then, the simulated rTMS was administered using a NeuroStar sham coil, which looked the same as the active stimulation coil and produced discharge noise and vibration without stimulating the cerebral cortex. This technique has been suggested to provide the most effective blinding compared to other methods used in randomized, controlled rTMS studies. The physician who set up the active and sham coils played no role in outcome measure assessments in order to maintain blinding.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
score on a scale
  Before rTMS | 17 (3.95) | 16.6 (4.92)
  Immediately after rTMS | 17 (5.35) | 15.8 (3.46)
  2 weeks after rTMS | 15.8 (4.78) | 16.3 (4.41)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Null hypothesis is that there was no interaction between the intervention and time factors on the TWSTRS scores; Test type: Superiority; p = 0.691, ANOVA; Two-way repeated measures ANOVA

2. Secondary Outcome: Beck Depression Inventory (BDI)
Description: This is a 21-question survey evaluating depression in patients on a 0 to 3 scale, with a minimum score of 0 and maximum score 63, and higher score indicating a higher level of depression.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active rTMS: The active or sham repetitive transcranial magnetic stimulation (rTMS) was provided at 9 weeks following the botulinum toxin injection.
  First, a clinical therapeutic NeuroStar TMS coil (Neuronetics, Malvern, PA) was used to determine the resting motor threshold (RMT), defined as the lowest stimulation intensity required to evoke a muscle twitch in a target muscle (first dorsal interosseus) for 5/10 pulses. The dPMC target was defined as 1 cm medial and 2 cm anterior to the site of RMT acquisition, consistent with how this target has been defined in the literature previously.
  Then, the clinical therapeutic TMS coil was switched to the active NeuroStar TMS coil. The rTMS protocol was as follows: each session consisted of 1-Hz rTMS over the dPMC for 30 minutes (1800 pulses) at 90% of the RMT. This study used an accelerated protocol: patients received 4 sessions per day for 4 consecutive days with a 10-minute break between each session. The daily duration of the rTMS protocol, including breaks, lasted approximately 160 minutes.
- Sham rTMS: The active or sham rTMS was provided at 9 weeks following the botulinum toxin injection.
  First, the participants underwent the same procedure for identifying the target location and RMT as was used in patients receiving active rTMS.
  Then, the simulated rTMS was administered using a NeuroStar sham coil, which looked the same as the active stimulation coil and produced discharge noise and vibration without stimulating the cerebral cortex. This technique has been suggested to provide the most effective blinding compared to other methods used in randomized, controlled rTMS studies. The physician who set up the active and sham coils played no role in outcome measure assessments in order to maintain blinding.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
score on a scale
  Before rTMS | 6.4 (6.39) | 8 (7)
  Immediately after rTMS | 4.8 (4.44) | 7.4 (4.83)
  2 weeks after rTMS | 6.4 (5.68) | 7.6 (6.02)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Null hypothesis is that there was no interaction between the intervention and time factors on the BDI scores; Test type: Superiority; p = 0.816, ANOVA; Two-way repeated measures ANOVA

3. Secondary Outcome: Trail-Making Test: Part A
Description: Patients are instructed to connect circles in ascending numerical order and are scored on how quickly they are able to complete the task. A longer amount of time indicates more severe cognitive impairment (in general, more than 78 seconds to complete Part A is considered impaired).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
seconds
  Before rTMS | 30.52 (9.78) | 28.92 (12.19)
  Immediately after rTMS | 24.77 (9.07) | 28.66 (12.27)
  2 weeks after rTMS | 25.97 (7.90) | 22.26 (5.69)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Null hypothesis is that there was no interaction between the intervention and time factors on the time to complete the TMT-A task; Test type: Superiority; p = 0.167, ANOVA; Two-way repeated measures ANOVA

4. Secondary Outcome: Trail-Making Test: Part B
Description: Patients are instructed to connect circles in ascending numerical order and are scored on how quickly they are able to complete the task. A longer amount of time indicates more severe cognitive impairment (in general, more than 273 seconds to complete Part B is considered impaired).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
seconds
  Before rTMS | 72.70 (46.08) | 72.77 (49.14)
  Immediately after rTMS | 73.88 (31.98) | 66.44 (50.40)
  2 weeks after rTMS | 60.28 (29.38) | 68.48 (48.29)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.507, ANOVA; Two-way repeated measures ANOVA

5. Secondary Outcome: Wisconsin Card Sorting Task (WCST) - %Total Errors
Description: The Wisconsin Card Sorting Test is a test of rule-learning and conceptual flexibility. The participant is required to learn to sort a series of cards according to one of three principles (color, form or number) based on response feedback. This measure is computed by calculating the ration of total errors to trials administered and multiplied by 100.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
percentage
  Before rTMS | 35.67 (15.57) | 25.25 (10.10)
  Immediately after rTMS | 36.98 (25.23) | 28.11 (20.49)
  2 weeks after rTMS | 25.52 (10.66) | 36.89 (27.75)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Superiority; p = 0.056, ANOVA; Two-way repeated measures ANOVA

6. Secondary Outcome: Wisconsin Card Sorting Task (WCST) - %Perseverative Errors
Description: The Wisconsin Card Sorting Test is a test of rule-learning and conceptual flexibility. The participant is required to learn to sort a series of cards according to one of three principles (color, form or number) based on response feedback. This measure reflects the "density" of perseverative errors in relation to the overall test performance. It is computed by calculating the ration of total errors to trials administered and multiplied by 100.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 5 | 5
percentage
  Before rTMS | 16.57 (11.92) | 15.30 (5.19)
  Immediately after rTMS | 15.76 (20.43) | 19.88 (15.44)
  2 weeks after rTMS | 16.39 (9.95) | 13.65 (13.72)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Superiority; p = 0.646, ANOVA; Two-way repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: All-Cause Mortality Serious Adverse Events Other Adverse Events
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=5) | Sham rTMS (N=5)
Headache (Nervous system disorders) | 1 (3) | 2 (2)
Neck discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04916444/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT04916444/SAP_003.pdf
  • Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT04916444/ICF_001.pdf